CLINICAL TRIAL: NCT02291601
Title: Assessment of the Antimicrobial Efficacy of 2% CHG Cloth Preoperative Skin Preparation
Brief Title: Preoperative CHG Cloth on Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R13-052
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Surgery
Keywords: Preoperative surgical skin preparation
MeSH Terms: interventions — chlorhexidine gluconate; Chromogranins; Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine Gluconate Cloth (Experimental): 2% CHG, single application
  Interventions: Drug: Chlorhexidine Gluconate
- Vehicle Cloth (Placebo Comparator): Excipients on cloth
  Interventions: Other: Vehicle
- Active Chlorhexidine gluconate solution (Active Comparator): Dynahex 2% CHG
  Interventions: Drug: DynaHex-2

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — comparison with other CHG products
  Other Names: CHG
  Arms: Chlorhexidine Gluconate Cloth
Other: Vehicle — Excipients of CHG product only.
  Other Names: Control
  Arms: Vehicle Cloth
Drug: DynaHex-2 — 2% CHG solution
  Other Names: CHG 2% Solution
  Arms: Active Chlorhexidine gluconate solution

SUMMARY:
Evaluate the effects of CHG cloth on the reduction of bacteria on the skin.

DETAILED DESCRIPTION:
Examine the antimicrobial cloth effects on normal flora bacteria of the abdomen and groin area post CHG application.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females
* 16 years of age or older
* Signed informed consent
* Good Health
* Six inches of abdomen and groin areas without tattoos, or skin disorders

Exclusion Criteria:

* Dermatological Conditions
* Sensitivity to latex
* Sensitivity to CHG

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C Beausoleil, Principal Investigator — BS
Locations (1):
- BioScience, Butte, Montana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared with FDA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon achieving sufficient microbial growth prior to product application on either the abdomen, groin or both abdomen and groin regions, sites of the participant were then randomized to receive one or two products for evaluation for up 4 sites. Differences in the number of participants is based on microbial qualification.
Pre-assignment Details: The sites of the participant were tested for microbial activity after product application. In some instances, more than one product could have been applied to a participant but only one product per site (groin and/or abdomen sites). Up to 4 sites could be treated : 1) both groin and abdomen, 2) only the groin or 3) only the abdomen.
Units Other Than Participants: sites
Groups:
- CHG Cloth: CHG 3 min application
- Vehicle: Vehicle, 3 min application
- Comparator CHG: marketed CHG - application done per products instructions for use
Period: Abdomen
Arm/Group | CHG Cloth | Vehicle | Comparator CHG
Started | 638; 638 sites | 108; 108 sites | 642; 642 sites
Completed (Completed is a lower participant number than started due to failed treatment day baselines) | 305; 305 sites (638 participants received CHG cloth) | 54; 54 sites (108 participants received vehicle) | 303; 303 sites (642 participants received comparator CHG)
Not Completed | 333; 333 sites | 54; 54 sites | 339; 339 sites
Not completed — Did not qualify | 333 | 54 | 339
Period: Groin
Arm/Group | CHG Cloth | Vehicle | Comparator CHG
Started | 520; 520 sites | 93; 93 sites | 515; 515 sites
Completed (Completed is a lower participant number than started due to failed treatment day baselines) | 337; 337 sites (520 participants received CHG cloth) | 63; 63 sites (93 participants received vehicle) | 338; 338 sites (515 participants received Comparator CHG)
Not Completed | 183; 183 sites | 30; 30 sites | 177; 177 sites
Not completed — Did not qualify | 183 | 30 | 177

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants represents the total number of participants that qualified and were tested.
Groups:
- CHG, Vehicle, Comparator CHG: Single applications of products. 3 min application for CHG and vehicle. Comparator CHG applied according to instructions.
Arm/Group | CHG, Vehicle, Comparator CHG
Number analyzed (Participants) | 879
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 829
  >=65 years | 37
Age, Continuous [Mean (Full Range); unit: years] | 35 [16 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281
  Male | 598
Region of Enrollment [Number; unit: participants]
  United States | 879

OUTCOME MEASURES:

1. Primary Outcome: Percent Responder Rates of Bacterial Reduction on the Abdomen and Groin Sites
Description: Percent of abdomen and groin sites that achieve a 2-Log or 3-Log reduction respectively of bacterial flora from baseline.
  Note: The number of participants in each treatment group (abdomen and/or groin) can vary depending on whether participants achieved qualifying microbial levels on the abdomen and groin at baseline.
Time Frame: 10 minutes to 8 hours
Population: Participants received 1 or 2 products on up to 2 abdomen and 2 groin sites, 2 abdomen only sites or 2 groin sites only.
Measure: Number; unit: % of Treated Sites
Units Other Than Participants: sites
Groups:
- CHG Abdomen; Vehicle Abdomen; Comparator Abdomen: single application on abdomen
- CHG Groin; Vehicle Groin: single application on groin.
- Comparator Groin: single application of groin
Arm/Group | CHG Abdomen | CHG Groin | Vehicle Abdomen | Vehicle Groin | Comparator Abdomen | Comparator Groin
Number analyzed (Participants) | 305 | 337 | 54 | 60 | 303 | 338
Number analyzed (sites) | 305 | 337 | 54 | 60 | 303 | 338
% of Treated Sites
  10 min | 80 | 75 | 86 | 65 | 81 | 68
  6 hours | 99 | 100 | 97 | 100 | 96 | 100
  8 hours | 98 | 100 | 97 | 100 | 96 | 100

ADVERSE EVENTS:
Description: Qualified and disqualified participants were included in the safety analysis for each treatment group as all of these participants were exposed to one or two different products. In those cases where one participant received 2 products at the same time (on different sites), participants were represented for both products.
Groups:
- CHG Cloth: single application
- Comparator CHG: 2% CHG solution
Arm/Group | CHG Cloth | Vehicle | Comparator CHG
Serious Adverse Events (participants affected / at risk) | 0/755 | 0/136 | 0/753
Other Adverse Events (participants affected / at risk) | 16/755 | 4/136 | 8/753
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHG Cloth (N=755) | Vehicle (N=136) | Comparator CHG (N=753)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1) | 3 (3)
Irritation skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (5) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential information based on contract